CLINICAL TRIAL: NCT05721573
Title: A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of ABC008 in the Treatment of Subjects With Inclusion Body Myositis
Brief Title: A Study to Evaluate the Efficacy and Safety of ABC008 for Inclusion Body Myositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abcuro, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC008-IBM-201
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Inclusion Body Myositis
Keywords: Muscular Diseases; Inflammatory Myopathy; Myositis; Neuromuscular Diseases; Nervous System Disease
MeSH Terms: conditions — Myositis, Inclusion Body; Muscular Diseases; Myositis; Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 mg/kg ABC008 (Active Comparator): Part A - ABC008 N=12
  Part B - ABC008 N= 67
  Interventions: Drug: ABC008
- 2.0 mg/kg ABC008 (Active Comparator): Part A - ABC008 N=12
  Part B - ABC008 N= 67
  Interventions: Drug: ABC008
- Placebo (Placebo Comparator): Part A - Placebo N= 6
  Part B - Placebo N= 67
  Interventions: Drug: ABC008

INTERVENTIONS:
Drug: ABC008 — Given by subcutaneous injection

SUMMARY:
A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Determine the Efficacy and Safety of ABC008 in the Treatment of Subjects with Inclusion Body Myositis

DETAILED DESCRIPTION:
A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Determine the Efficacy and Safety of ABC008 in the Treatment of Subjects with Inclusion Body Myositis Detailed Description: A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Determine the Efficacy and Safety of ABC008 in the Treatment of Subjects with Inclusion Body Myositis Detailed Description: This is a Phase II/III randomized, double-blind, placebo-controlled, parallel multicenter study with 3 parts.

The study will include a sentinel cohort (Part A) of 30 subjects who will receive first three doses of the study drug. Safety data from subjects in the sentinel cohorts will be evaluated by a Data and Safety Monitoring Board (DSMB) before further dosing of the sentinel cohort, as well as initiation of enrollment in the double-blind safety and efficacy cohort (Part B). After completion of Part A or Part B, subjects have the option of enrolling in an open-label long-term extension study or progressing to the pharmacodynamics (PD) recovery cohort (Part C), to evaluate the recovery of the depletion of killer cell lectin-like receptor G1 (KLRG1)+ cells after the end of treatment with ABC008.

Efficacy, safety, HRQoL, and HRU assessments will be conducted. Blood samples will be obtained to evaluate the serum PK, PD, and immunogenicity of ABC008 throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females age >40 years at the time of the first dose of study medication;
* Weight >40 and <150 kg;
* Diagnosis of either clinico-pathologically defined IBM, clinically defined IBM, or probable IBM according to the European Neuromuscular Centre (ENMC) IBM 2011 research diagnostic criteria (Rose et al., 2013). Documented histopathology results must be available prior to Baseline (Day 1) to confirm eligibility;
* Able to arise from a chair (with armrests), with use of their arms but without support from another person or device (e.g., cane, walking stick), at Screening and Baseline (Day 1);
* Able to walk 3 meters, turn around, walk back to the chair, and sit down, with or without assistive device. Once arisen from the chair, subject may use any walking device but cannot be supported by another person, furniture, or a wall;

Exclusion Criteria:

* Any other form of myositis or myopathy other than IBM, e.g., metabolic or drug-induced myopathy, drug-induced myositis, anti-synthetase syndrome, polymyositis or dermatomyositis, cancer-associated myositis (myositis diagnosed within 3 years, either before or after), myositis in overlap with another autoimmune disease (e.g., systemic lupus, systemic sclerosis, rheumatoid arthritis), or muscular dystrophy;
* Any condition, e.g., severe degenerative arthritis with limited range of motion, which precludes the ability to quantitate muscle strength or perform functional assessments (e.g., mTUG), in the Investigator's opinion;.
* Presence of another autoimmune or autoinflammatory disease other than indication under study, e.g., rheumatoid arthritis, psoriatic arthritis, axial spondyloarthropathy, inflammatory bowel disease, systemic lupus erythematosus. Subjects with Sjogren's syndrome, T-cell large granular lymphocyte leukemia (T-LGLL), or well-controlled thyroid disease are permitted;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Part A - To determine the safety and tolerability of recurrent dosing of ABC008 in subjects with IBM at 2 SC dose levels. | From Baseline (week 0) through week 20.
  Safety as assessed by the incidence, type and severity of Treatment Emergent Adverse Events (TEAEs)
Part B - To determine the efficacy of ABC008 in IBM at two SC dose levels as measured by IBM Functional Rating Scale (IBMFRS) at Week (W)76 | From Baseline (week 0) through study completion, an average of 76 weeks
  Mean change in IBM Functional Rating Scale (IBMFRS)

SECONDARY OUTCOMES:
Part A - Treatment Emergent Serious Adverse Events (TEASAEs) | From Baseline (Day 1) through study completion, an average of 80 weeks.
  Incidence, type and severity of TEASAEs.
Part A - Treatment Emergent Adverse Events (TEAEs) onset within 24 hours of Study Medication Administration. | From Baseline (Day 1) through study completion, an average of 80 weeks.
  Incidence, type, and severity of TEAEs with onset within 24 hours from the start of any of study medication administration
Part A - Treatment Emergent Adverse Events leading to study medication or study discontinuation. | From Baseline (Day 1) through study completion, an average of 80 weeks.
  Incidence of TEAEs leading to study medication or study discontinuation
Part A - Clinically significant changes in standard laboratory parameters, vital signs, and ECGs | From Baseline (Day 1) through study completion, an average of 80 weeks.
  Incidence of clinically significant changes in standard laboratory parameters, vital signs, and ECGs
Part A - Adverse Events of Special Interest (AESI) | From Baseline (Day 1) through study completion, an average of 80 weeks.
  Incidence of AESIs.
Part B - Manual Muscle Test 12 (MMT 12) | From Baseline (Day 1) through study completion, an average of 76 weeks.
  Mean change in MMT 12
Part B - Hand Grip Dynamometry | From Baseline (Day 1) through study completion, an average of 76 weeks.
  Mean change in hand grip strength by dynamometry.
Part B - Quadriceps Dynamometry | From Baseline (Day 1) through study completion, an average of 76 weeks.
  Mean change in quadriceps strength by dynamometry.
Part B - Modified Timed Up and Go (mTUG) | From Baseline (Day 1) through study completion, an average of 76 weeks.
  Mean change in mTUG.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (34):
  - Neuromuscular Research Center, Phoenix, Arizona
  - University of California Irvine Medical Center (UCIMC) - Amyotrophic Lateral Sclerosis (ALS) and Neuromuscular Center, Irvine, California
  - Keck Hosptial of USC, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Neuroscience Medical Center, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Hospital Anschutz Outpatient Pavillion, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Memorial Hospital, Department of Neurology (Clinic), Chicago, Illinois
  - University of Kansas Medical, Kansas City, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Neuromuscular Diagnostic Center - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center / The Neurological Institute of New York, New York, New York
  - Duke Neurological Disorders Clinic -1L, Durham, North Carolina
  - Wake Forrest School of Medicine, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Arthritis and Autoimmunity Center, Falk Clinic, Pittsburgh, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Texas Neurology, Dallas, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Virginia Commonwealth University, Henrico, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- AZ Sint-Lucas & Volkskliniek, Ghent, Belgium
- Canada (2):
  - Heritage Medical Research Clinic - University of Calgary, Calgary, Alberta
  - Genge Partners Inc., Montreal, Quebec
- Hospital Pitie-Salpetriere - AP-HP, Paris, France
- Germany (2):
  - Krankenhaus und Poliklinik Rüdersdorf GmbH, Berlin
  - University Hosptial Duesseldorf, Düsseldorf
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, National Hospital for Neurology and Neurosurgery (NHNN), London
  - Salford Royal Hospital, Northern Care Alliance NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — http://abcuro.com